CLINICAL TRIAL: NCT04701242
Title: Ezetimibe Utilization Early After Acute Myocardial Infarction. "EzAMI Trial"
Brief Title: Ezetimibe Utilization Early After Acute Myocardial Infarction, "EzAMI Trial"
Acronym: EzAMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Aswan Heart Centre (Other)
Responsible Party: Principal Investigator, Ahmad Samir, Lecturer of Cardiology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20200902MYFAHC_EzAMI
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Acute Myocardial Infarction; Dyslipidemias
Keywords: Statin failure, acute myocardial infarction, ezetimibe
MeSH Terms: conditions — Dyslipidemias | interventions — Ezetimibe

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized controlled trial 1:1 randomization
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will receive blinded drug containers. Care providers and investigators assessing study end-points will be blinded to group allocation of the patients Steering committee will be the only who have the key table for study-ID of the patient and allocation groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin-Ezetimibe combination (Active Comparator): Eligible patients randomized to this arm will receive combination of Atorvastatin 80mg plus Ezetimibe 10mg
  Interventions: Drug: Ezetimibe 10mg
- Atorvastatin monotherapy (No Intervention): Eligible patients randomized to this arm will receive Atorvastatin 80mg as monotherapy for LDL-C reduction. They can be upgraded to combination (adding Ezetimibe 10mg) if found in follow-up that they had not achieve recommended LDL-C targets.

INTERVENTIONS:
Drug: Ezetimibe 10mg — comparing upfront use of Ezetimibe (added to high intensity statins) after acute myocardial infarction versus selective Ezetimibe initiation to those failing to achieve LDL-C targets when assessed in follow up visit.
  Arms: Atorvastatin-Ezetimibe combination

SUMMARY:
Rationale:

Patients with acute coronary syndromes are at an increased risk for recurrent adverse coronary events, particularly during the early period following their initial presentation. Early (in-hospital) initiation of high-intensity statins reduces the risk of recurrent events and is therefore recommended by the best current practice guidelines.(1,2) However, the delayed onset of action of statin therapy and given the frequent failure of patients to achieve the recommended LDL-C targets using statins alone (as per the current practice guidelines recommendations), might be placing large number of patients at increased risk during such a vulnerable period early after an ACS.(3) More rapid and effective reduction of LDL-C levels using combination therapy from the outset may therefore be beneficial in these patients. This hypothesis has been tested with combining Evolocumab and a statin in the recent EVOPACS study, in which this combination after ACS has shown to be safe and more effective in achieving LDL-C targets at 6 weeks compared to statin monotherapy.(4) However, Evolocumab (a PCSK9i) is an expensive drug which is not affordable by many healthcare systems in low- and middle-income countries. Ezetemibe, on the other hand, is a safe and a cheap drug that can prove to be extremely cost-effective if a meaningful and timely reduction in LDL-C levels can be achieved when combined with a statin early after an ACS.

Study population Patients presenting with acute myocardial infarction, with baseline LDL-C levels not likely to achieve recommended targets on statin monotherapy. This is assumed to be with LDL-C level > 125 mg/dl for those not on lipid lowering therapy; or with LDL-C > 100 mg/dl on moderate intensity statin therapy at the time of presentation.

Study design Prospective randomized controlled single-blinded trial. A sample size of 500 patients, 250 in each arm, was calculated to provide a power of 0.9 and an adjusted type 1 error as 0.05.

Primary outcomes

* Percentage of patients achieving target LDL-C levels (<70 mg/dl) at 6 weeks interval. (Efficacy endpoint)
* Freedom from alanine transaminase elevation (ALT) more than 3 folds upper reference limit "URL" or statin associated muscle symptoms associated with CK elevation more than 4 folds URL. (Safety endpoint) Secondary outcomes
* Percentage of patients achieving > 50% reduction of LDL-C and to levels below 70mg/dl at 6 weeks interval.
* Percentage of LDL-C reduction at 6 weeks interval.
* Reduction of high-sensitive C-reactive protein (hs-CRP) from baseline to 6 weeks interval.
* Correlating statins efficacy to reduce LDL-C and likelihood to cause statins related adverse effects to genetic alleles of ABC [ATP Binding Cassette] types A1, G5 and G8, and of CYP450 isoenzymes.
* MACE free survival at 1 year, (CV death; non fatal-MI; hospitalization for ACS, urgent unplanned revascularization and stroke).

DETAILED DESCRIPTION:
Introduction:

After a major event of "atherosclerotic cardiovascular disease" ASCVD, like a stroke or "Acute Myocardial infarction" AMI, best practice clinical guidelines strongly recommend prompt initiation of high-intensity statin therapy for secondary prevention of recurrent events.1-4 Owing to its plaque stabilization effects, pleotropic anti-inflammatory effects, besides its "Low Density Lipoprotein-Cholesterol" LDL-C lowering effects, statins received the highest levels of recommendations in these settings.5,6 We learnt from the Cholesterol Treatment Trialist "CTT" collaboration through studying 170,000 cases from 26 trials, that the magnitude of LDL-C reduction is translated into a proportionate reduction of adverse events.7 It was found that every 1 mmol/L (38.8 mg/dl) reduction in LDL-C is paralleled by a 22% in major vascular events (AMI-death- stroke- any revascularization); 23% in major adverse coronary events; 20% in coronary artery disease deaths; 17% in total stroke and by 10% in total deaths.7 Hence, in secondary prevention of ASCVD, guidelines clearly instructs for aggressive reduction of LDL-C by at least 50% of baseline values and to levels <70 mg/dl or <55 mg/dl for ACC or ESC guidelines respectively.1,2 Nevertheless, both guidelines instructed to initiate statins monotherapy after the index event, and to add other agents (mainly; Ezetimibe or PCSK9i) if targets were found not have been achieved in follow-ups.1,2 High intensity statins as monotherapy are expected according to ESC and ACC guidelines1,2 to reduce LDL-C levels by about 50%, while according to the NICE guidelines4 by 40%. However, most reports from real life experience quite often revealed no more than 35%-to-40% reductions.8,9 Thus, failures to achieve target LDL-C levels is quite prevalent, and obviously is more common with higher baseline LDL-C levels. In the data published from the PINNACLE registry involving 1.9 million patients with ASCVD, only 31.9% of those on statin monotherapy could achieve LDL-C <70 mg/dl.10 Similar results were reported in the NHANES, EUROASPIRE and GOULD registries.8,11,12 There is large body of evidence that the early period after an ASCVD event is the most vulnerable period for recurrent events.7,13,14 The previously mentioned benefits in CTT were observed over 5 years of follow-up, yet, the magnitude of risk reduction in the earliest 12 months was equal to the cumulative reduction in the subsequent 4 years.7 In a sub-analysis from the FOURIER trial, intensifying LDL-C reduction by combining Evolocumab with maximum tolerated statins resulted in larger risk reduction in those with recent (≤12 months) MI compared to those with remote (>12 months) MI; with a RRR for CV death, MI or stroke of 25% vs 15%).15 Plausibly, the absolute benefit of intensified preventive measures is maximized when the absolute risk is more. It can be arguable that initiating combination LDL-C lowering therapies promptly after AMI would be more appropriate than endangering more than two thirds of the patients who would fail to achieve LDL-C targets through such a vulnerable period awaiting to establish the indication in follow-up visits. This is of particular concern in patients with high baseline LDL-C expected not to achieve goals with statins alone.1,2 The EVOPACS study, "Evolocumab for Early Reduction of LDL-Cholesterol Levels in Patients with Acute Coronary Syndromes" tested atorvastatin 40 mg alone compared to combining atorvastatin 40 mg plus PCSK9 Evolocumab 420 mg started during index hospitalization and repeated after 4 weeks.9 At 8 weeks interval, LDL-C was reduced by 35.4% in the atorvastatin group compared to 77.1% in Evolocumab + atorvastatin (from 3.42±0.94 mmol/L to 2.06±0.63 and from 3.61±1.00 mmol/L to 0.79±0.46 respectively). Worth mentioning that by the 8 weeks follow up time, achieving LDL-C < 70 mg/dl (1.8 mmol/L) occurred only in 37.6% in the statin monotherapy compared to 95.7% in the combination arm.9 Despite the high potency of PCSK9 inhibitors in LDL-C reduction, the ACC describes them as overpriced and not cost-effective in the contemporary prices.2 Ezetimibe is a very affordable agent that inhibits exogenous cholesterol absorption by acting on Nieman-pick C1 like1 protein. It is a safe and well tolerated drug that need no dose reduction or adjustment in moderate renal or hepatic dysfunction. Because of acting at different hinge points, Ezetimibe acts additively to statins and leads to further 20% reduction of serum LDL-C levels.16,17 The current ACC 2018 guidelines for cholesterol management gave a class (I) level of evidence (B) that patients with ASCVD judged to be at very high risk and are considered for PCSK9 inhibitors, should be receiving maximally tolerated statins and ezetimibe.2 In the IMPROVE-IT, "IMProved Reduction of Outcomes: Vytorin Efficacy International Trial", adding Ezetimibe to Simvastatin 40 mg reduced MACE by 6.4% compared to Simvastatin 40 mg alone in patients with ACS and LDL-C > 125 mg/dl.17 Though such results are in favor of combining Ezetimibe with statins after ACS, yet Simvastatin at the dose of 40 mg is a moderate intensity statin and up titration to 80 mg is strongly discouraged.1,2 Moreover, Simvastatin is characterized by multiple drug-drug interactions, an issue that increased chances for side effects, intolerance and thus treatment discontinuation compared to the currently more often used atorvastatin and rusovastatin.2,16 Being safe and affordable, upfront combination of high intensity statin plus ezetimibe to AMI patients might be more effective in achieving LDL-C targets and reducing adverse events compared to the current practice of initiating statin monotherapy and deferring intensification weeks-to-months till the time of follow-up.

Aim of the Work Evaluate safety and efficacy of initiating combined ezetimibe plus statin therapy compared to statin monotherapy early after AMI.

Ethical Considerations The study shall be launched after ethical committee approval. Informed consents will be obtained from eligible participants prior enrollment to the study. Patients will be fully oriented about the benefits and potential adverse effects by participation. They will be given a shortcut access (through the study team direct contact) in cases any problems or complaints occurred. Possible side effects of any of the used medications will be thoroughly discussed with the patients for early identification and swift reporting to the research team. Patients will be informed about the schedule of follow up visits and about the study-dictated laboratory workup. Patients' identity and data are completely confidential and will not be disclosed except to treating physicians. All clinical, laboratory data and data from genetic tests will be dealt with complete confidentiality. Data for analysis and laboratory results will be anonymized before they are given to the statistical team, and thus study results will be devoid of any personal data.

Methodology I. Study design A Prospective Randomized Controlled Study. II. Study setting and location The study will be conducted in and fully supported by Aswan Heart Centre, Magdi Yacoub Foundation.

The researchers do not have any connections to industry, did not (and will not) receive funds or support from any sponsors.

III. Study population Patients presenting by acute myocardial infarction, (both STEMI and NSTEMI are included). Diagnosis will depend on clinical presentation, twelve-lead ECG, cardiac biomarkers and echocardiography when diagnosis is doubtful as recommended by the 4th universal definition of myocardial infarction.18 IV. Eligibility Criteria Patients presenting by AMI who are likely not to achieve LDL-C targets on statin monotherapy.

1. Inclusion criteria

* Age more than 18 years. Both genders are eligible.
* Acute myocardial infarction (STEMI or NSTEMI) within 48 hours from the onset of symptoms.
* Baseline LDL-C above 125 mg/dl for those who were not on consistent lipid lowering therapy; or above 100 mg/dl for those who were compliant (≥ 90 days) on moderate intensity statin therapy.

  2. Exclusion criteria
* Refusal to participate in the study.
* Proved intolerance to statins on previous use.
* Having conditions (or taking medications) that would not allow concomitant safe statins use. [such as patients receiving Cyclosporine - Gemfibrozil -Pazopanib - Tipranavir - Itraconazole - Ketoconazole]
* Those who are already compliant on high intensity statins.
* Those who are already on statins plus non-statin agent (ezetimibe-PCSK9i-BAS).
* Known familial dyslipidemia or having TG>500 mg/dl or LDL-C>190 mg/dl which are highly suggestive of familial or secondary causes.
* Pregnant or contemplating pregnancy in the following 12 months. [relevant for females in the child-bearing period] V. Study Procedures

  1. Randomization Within 48 hours of the onset of symptoms, a computer-generated sequence will be used for randomization into 1:1 fashion to allocate eligible patients into either; statin monotherapy (will receive atorvastatin 80 mg) or statins-ezetimibe combination (will receive atorvastatin 80 mg + ezetimibe 10 mg).
  2. Study Protocol A baseline lipid profile will be checked within 48 hours from the AMI onset. A fasting lipid profile will be ordered if the triglycerides were > 400 mg/dl in the non-fasting results. Eligible patients will be recruited after explaining the study protocol and acquiring a written informed consent. A venous blood sample for genetic analysis will be provided to perform cutting edge next generation sequencing to investigate for genetic alleles of ATP Binding Cassette (ABC) types A1, G5, G8 and CYP450 and correlate isoform variants with statins responsiveness and efficacy to achieve LDL-C targets. Genetic sequencing will be performed using high throughput sequencers.

Management of the AMI will be according to the most recent guidelines' recommendations including both the interventional and the medical aspects. The statin monotherapy arm will receive atorvastatin 80 mg once daily as their lipid lowering therapy, compared to the combination therapy arm who will receive atorvastatin 80 mg plus ezetimibe 10 mg once daily. To ensure blinding and compliance, participants will be provided free of charge with 2 differently colored packings for lipid control through the 12 months of the study. In the statins alone arm both will contain atorvastatin 40mg tablets, while for the combination arm one of them will contain atorvastatin/ezetimibe 40/10mg and the other will be atorvastatin 40mg tablets. Patients will be instructed to have 1 tablet from each packing at night.

Apart from LDL-C management, life-style interventions and all other guidelines directed medical therapy (GDMT) will be equally implemented in both arms. The study team, as part of the general practice in AHC, will be consolidating advices for compliance to life-style interventions and all other GDMT, but will not be providing them.

Hs-CRP, ALT, CK and lipid profile will be tested at baseline and at 6 weeks of the study. Repeating these or ordering any other laboratory workup will be allowed at any other time deemed clinically indicated. Patients on the statin monotherapy arm not achieving target LDL-C levels on the 6-weeks follow-up will be prescribed ezetimibe in addition to their regimen (as per current best practice guidelines) but will remain labelled as initial monotherapy group.

Participants will have a clinical follow-up visit at 6 weeks, 6 months then at 1 year. However, they will be instructed to contact the research team at any relevant clinical complaint or emergency. Magdi Yacoub foundation is completely responsible for the management of any clinical complication or adverse events resulting from (or related to) the study agent. After the study ends (1 year), participants will be offered the regular follow-up appointments according to AHC institutional policy.

VI. Study outcomes

1. Primary outcome

   * Percent of patients who achieve required LDL-C targets according to the ACC guidelines (<70 mg/dl) at 6 weeks interval. (Efficacy endpoint)
   * Freedom from Alanine Transaminase elevation (ALT) more than 3 folds upper reference limit OR muscle pains associated with CK elevation more than 4 folds upper reference limit. (Safety endpoint)
2. Secondary outcomes

   * Percent of patients achieving > 50% reduction from baseline and to a level <70 mg/dl of LDL-C to 6 weeks interval.
   * Percent of LDL-C reduction from baseline to 6 weeks interval.
   * Reduction of high-sensitive C-reactive protein (hs-CRP) from baseline to 6 weeks interval.
   * Correlating efficacy of statins to reduce LDL-C and/or cause statins related adverse effects to genetic alleles of ABC types A1, G5 and G8 and CYP450 which are believed to impact statins pharmacokinetics and pharmacodynamics.
   * MACE free survival at 1 year, (cardiovascular death; non fatal-MI; hospitalization for ACS, urgent unplanned revascularization, and cerebrovascular stroke).

Statistical Analysis I. Sample size Sample size was calculated using MedCalc Statistical Software version 19.0.4 (MedCalc Software, Ostend, Belgium; https://www.medcalc.org; 2019) adjusting margin for type 1 error as 0.05 and utilizing a study power of 90%. The expected proportion of patients on statin monotherapy achieving LDL-C targets was adjusted to 50% (it was 37.6% in the control arm of EVOPACS 9) and we expected that this proportion to be 70% in the combination group. Accordingly, a minimum sample of 268 patients randomized in 1:1 fashion was suggested. The research group planned to have a sample of 500 patients on 2 groups of 250 each.

II. Statistical analysis Statistical package for social science (SPSS) software, version 22 for Microsoft Windows (SPSS Inc., Chicago, IL, USA) will be used for data analysis. Categorical data will be presented as frequency and percentages (n (%)) and correlations among them will be analysed by chi square test. Continuous data will be checked for normality using Shapiro-Wilk test and will be presented as mean (standard deviation) or median (interquartile range) as appropriate. Continuous data will be analysed using one-way analysis of variance (ANOVA). Repeated measures will be analysed using analysis of variance (ANOVA) for repeated measures with post-hoc pairwise comparisons using the Tukey and Bonferroni tests. A probability p value less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years. Both genders are eligible.
* Acute myocardial infarction (STEMI or NSTEMI) within 48 hours from the onset of symptoms.
* Baseline LDL-C above 125 mg/dl for those who were not on consistent lipid lowering therapy; or above 100 mg/dl for those who were compliant (≥ 90 days) on moderate intensity statin therapy.

Exclusion Criteria:

* Refusal to participate in the study.
* Proved intolerance to statins on previous use.
* Having conditions (or taking medications) that would not allow concomitant safe statins use. [such as patients receiving Cyclosporine - Gemfibrozil -Pazopanib - Tipranavir - Itraconazole - Ketoconazole]
* Those who are already compliant on high intensity statins.
* Those who are already on statins plus non-statin agent (ezetimibe-PCSK9i-BAS).
* Known familial dyslipidemia or having TG>500 mg/dl or LDL-C>190 mg/dl which are highly suggestive of familial or secondary causes.
* Pregnant or contemplating pregnancy in the following 12 months. [relevant for females in the child-bearing period]

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint | Six weeks
  ● Percent of patients who achieve required LDL-C targets according to the ACC guidelines (<70 mg/dl) at 6 weeks interval.
(Safety endpoint) | Six weeks
  ● Freedom from Alanine Transaminase elevation (ALT) more than 3 folds upper reference limit OR muscle pains associated with CK elevation more than 4 folds upper reference limit.

SECONDARY OUTCOMES:
● Percent of LDL-C reduction from baseline to 6 weeks interval. | Six weeks
● Reduction of high-sensitive C-reactive protein (hs-CRP) from baseline to 6 weeks interval. | Six weeks
● MACE free survival at 1 year, (cardiovascular death; non fatal-MI; hospitalization for ACS, urgent unplanned revascularization, and cerebrovascular stroke) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Samir, MD, Principal Investigator — Cairo University
Locations (1):
- Aswan Heart Centre, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided